CLINICAL TRIAL: NCT04615520
Title: A Multicenter Comparison of Risk Prediction Tools for Emergency Laparotomy in Greece
Brief Title: Evaluation of Surgical Risk Prediction Tools.
Status: Completed | Type: Observational
Sponsor: University Hospital of Crete (Other)
Collaborators: Nicosia General Hospital (Other); Laikο General Hospital, Athens (Other); Attikon Hospital (Other); Evangelismos Hospital (Other); Trikala General Hospital, Trikala (Unknown); Ippokrateio General Hospital of Thessaloniki (Other); General Hospital of Volos (Other); General University Hospital of Patras (Other); University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Konstantinos Lasithiotakis, Adj Professor of Surgery, University Hospital of Crete
Other Study IDs: 1681/26-02-2020
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Emergency Laparotomy
Keywords: emergency laparotomy; risk prediction; postoperative mortality; NELA; ACS-risk calculator; POSSUM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: In modern surgery, the prediction of perioperative death gains significant importance due to the availability of treatment options, means of improving the surgical outcome and for proper patient information. However, patient heterogeneity and the existence of multiple risk prediction tools complicate the prediction of perioperative mortality. Thus, prognostic tools are developed based on the analysis of preoperative variables. Most commonly used models are POSSUM, ACS-NSQIP, NELA and POTTER. The models have been assessed in West-European and North-American populations, each with different prognostic value.

Aim: Comparative analysis of predictive accuracy of the aforementioned risk prediction tools in Greek population.

Materials and Methods: The study is multicenter, non-interventional, prospective and observational and includes patients undergoing emergency laparotomies of general surgery. In cases of multiple operations in one hospitalization, the first operation is included. The clinical-laboratory variables, derived from POSSUM, NELA, ACS-NSQIP and POTTER models are recorded anonymously in a secure online database, REDCap (Research Electronic Data Capture).The minimum estimated number of included patients in order to accomplish statistically significant results is 600. Each of the centers submitted in the study, is expected to include approximately 60 patients in a period of 6-12 months. For the statistical analysis of data, Brier Score will be used and ROC with statistical significance lower than 0.05.

Conclusions: Upon completion of this study, the most accurate perioperative risk prediction tool in the Greek population is expected to be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18yrs
* Emergency laparotomy (operation simultaneously with resuscitation usually within one hour) or urgent (operation as soon as possible after resuscitation, within 24hrs)
* Operation in the gastrointestinal tract:
* Open or laparoscopic, or laparoscopically assisted procedures.
* Procedures involving the stomach, small or large bowel, or rectum for conditions such as perforation, ischaemia, abdominal abscess, bleeding or obstruction
* Wash out/evacuation of intraperitoneal abscess or haematoma
* Bowel resection/repair due to incarcerated/incisional hernias
* Bowel resection or repair due to incarcerated umbilical, inguinal or femoral hernias
* Open or laparoscopic adhesiolysis
* Laparotomy/laparoscopy with inoperable pathology
* Return to theatre for repair of a substantial dehiscence of major abdominal wound (i.e. "burst abdomen")
* Return to theatre after any operation (including vascular, gynecology, urology, cardiac) meeting the criteria above
* In the case of multiple procedures in the abdominopelvic cavity the patient is included if the main procedure is a general surgical one (i.e. if bowel resection happens during an open aneurysm repair it should not be included)
* Any intra-abdominal procedure not identifiable within exclusion criteria should be included.

Exclusion Criteria:

* Patients under 18
* Elective operation
* Diagnostic laparoscopy or laparotomy where no other procedure is performed (NB, if no procedure is performed due to inoperable pathology, then include)
* Appendicectomy with or without drainage of localized abscess
* Cholecystectomy with or without drainage of localized abscess
* Hernia repair without bowel resection
* Minor abdominal wound revision
* Vascular surgery
* Gynecological surgery - c-section - ruptured ectopic pregnancy
* Surgery relating to organ transplantation
* Removal of dialysis catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in a surgical department during a 12-month study period (May 1, 2020 - May 1, 2021 ).
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Number of deaths within 30 days from emergency laparotomy | 30 days after emergency laparotomy
  Patients who died of any cause within 30 days from emergency laparotomy

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Lasithiotakis, Principal Investigator — University Hospital of Heraklion
Locations (1):
- Department of Surgery, University Hospital of Heraklion, Heraklion, Greece

IPD SHARING:
Plan to Share IPD: No
No there is no plan to make IPD available to other researchers.

REFERENCES:
- [Derived] Kokkinakis S, Kritsotakis EI, Paterakis K, Karali GA, Malikides V, Kyprianou A, Papalexandraki M, Anastasiadis CS, Zoras O, Drakos N, Kehagias I, Kehagias D, Gouvas N, Kokkinos G, Pozotou I, Papatheodorou P, Frantzeskou K, Schizas D, Syllaios A, Palios IM, Nastos K, Perdikaris M, Michalopoulos NV, Margaris I, Lolis E, Dimopoulou G, Panagiotou D, Nikolaou V, Glantzounis GK, Pappas-Gogos G, Tepelenis K, Zacharioudakis G, Tsaramanidis S, Patsarikas I, Stylianidis G, Giannos G, Karanikas M, Kofina K, Markou M, Chrysos E, Lasithiotakis K. Prospective multicenter external validation of postoperative mortality prediction tools in patients undergoing emergency laparotomy. J Trauma Acute Care Surg. 2023 Jun 1;94(6):847-856. doi: 10.1097/TA.0000000000003904. Epub 2023 Feb 2. PMID 36726191